CLINICAL TRIAL: NCT03720990
Title: Smith-Lemli-Opitz Syndrome: A Pilot Study of Cholic Acid Supplementation
Brief Title: Smith-Lemli-Opitz Syndrome and Cholic Acid
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: University of Colorado, Denver (Other); Children's Hospital Medical Center, Cincinnati (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0464-18-FB
Record Dates: First submitted 2018-10-24; First posted 2018-10-26 (Actual); Results first posted 2023-12-13 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Smith-Lemli-Opitz Syndrome
Keywords: 7-Dehydrocholesterol reductase deficiency
MeSH Terms: conditions — Smith-Lemli-Opitz Syndrome | interventions — Cholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cholic acid (Experimental): Participants will be treated with cholic acid 10 mg/kg body weight.
  Interventions: Drug: Cholic Acid

INTERVENTIONS:
Drug: Cholic Acid — Participants will be treated with cholic acid for 8 weeks
  Other Names: Cholbam

SUMMARY:
The purpose of this study is to determine whether dietary cholic acid therapy benefits people with Smith-Lemli-Opitz syndrome (SLOS) by leading to an increase in plasma cholesterol and reduction in harmful cholesterol precursors. SLOS participants will be treated with dietary cholic acid for 8 weeks and plasma cholesterol and cholesterol precursor metabolites will be measured.

DETAILED DESCRIPTION:
People with SLOS have a deficiency of the 7-dehydrocholesterol reductase enzyme that makes cholesterol. Consequently, they exhibit deficient cholesterol levels and increased cholesterol precursor lipids, which are thought to be toxic. Cholesterol itself normally regulates the cholesterol synthesis pathway in the body and under conditions of low cholesterol seen in SLOS, more of the toxic cholesterol precursors are made. Since cholesterol is also necessary for production of bile acids in the liver, which help digest dietary cholesterol from the intestine, it is likely that low cholesterol levels in SLOS impairs bile acids from being made, which in turn prevents dietary cholesterol from being absorbed properly and contributes to the cholesterol deficiency seen in SLOS. Raising cholesterol in SLOS people by improving its absorption from the diet is expected to decrease the potentially toxic cholesterol precursor lipids, and both changes would be theoretically beneficial for SLOS people.

The objective of this study is to determine whether treatment with cholic acid (a major bile acid made in the body that improves fat absorption) will increase dietary absorption of cholesterol, reverse plasma cholesterol deficiency, and reduce harmful cholesterol precursor lipids. These changes would be favorable for SLOS people. To accomplish this objective, SLOS participants will be given dietary cholic acid (brand name Cholbam, manufactured by Retrophin) for 8 weeks and plasma cholesterol and its precursor lipids will be measured before and while taking the drug.

SLOS participants who are between 2 years and 25 years of age and are taking supplemental dietary cholesterol for at least 3 months will be enrolled. Participants must be clinically stable and able to travel to a study site. No change in supplemental dietary cholesterol intake will be allowed during the study, and dietary records will be obtained throughout the study.

To qualify for cholic acid therapy, participants must have plasma cholesterol ≤125 mg/dl before starting cholic acid. Participants will be treated with cholic acid for 8 weeks and will have blood specimens drawn at baseline (day 0), 4-weeks, 8-weeks and 12 weeks (4 weeks after stopping cholic acid therapy).

ELIGIBILITY:
Inclusion Criteria:

* Ages 2-25 years.
* Participants (or their parents/legally-authorized representative) must provide signed informed consent.
* Assent must be obtained from those participants ages 7-17 years who are intellectually capable of understanding this study.
* Diagnosis of SLOS based on clinical features and biochemical + genetic confirmation.
* Participants are capable of traveling to the STAIR study site.
* Fasting plasma cholesterol ≤125 mg/dL during the Qualification Phase must be established before starting cholic acid therapy.
* Clinically stable at the time of enrollment
* Participants must be on a constant dietary cholesterol intake for at least 3-months prior to treatment with cholic acid.
* Participants must agree to make no changes in cholesterol supplementation during the STAIR study.
* SLOS participants who are taking antioxidants will be included. Participants must agree to make no changes in the antioxidant dose during this study.
* For females of childbearing age (who have begun menstruating), a negative pregnancy test must be documented at the start of the study (week 0/ baseline) and at the end of cholic acid administration (week 8).

Exclusion Criteria:

* Participants are unable to provide signed informed consent and/or verbal assent.
* Participants have an unstable clinical condition that would prevent completion of the study. Medically unstable participants would include those with severe liver disease, complex birth defects such as severe heart disease or renal dysplasia, those with severe respiratory compromise requiring tracheostomy, or those who are not likely to survive longer than 1 year.
* Participants are taking drugs, nutraceuticals, probiotics or other compounds that are known or suspected to affect sterol metabolism.
* Participants have transaminase elevations (>3-fold above the reference range) at baseline.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2021-03-27 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen R Elias, MD, Study Chair — University of Colorado - Colorado Children's Hospital; William B Rizzo, MD, Principal Investigator — University of Nebraska
Locations (2):
- United States (2):
  - Colorado Children's Hospital, Aurora, Colorado
  - University of Nebraska Medical Center, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: Yes
All data will be de-identified and submitted to the Database of Genotypes and Phenotypes (dbGAP), according to NIH regulations.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available one year after completion of the study. Data will be available indefinitely.
Access Criteria: Data will be made available to everyone.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment conducted at Children's Hospital and Medical Center (CHMC), Omaha, NE and Childrens Hospital Colorado (CHCO).
Period: Overall Study
Arm/Group | Cholic Acid
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 12
Units Other Than Participants: plasma
Arm/Group | Cholic Acid
Number analyzed (Participants) | 12
Number analyzed (plasma) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 9.5 [2 to 27]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
Cholesterol [Count of Participants; unit: Participants] | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma Cholesterol
Description: Plasma cholesterol will be measured. Response to cholic acid treatment will consist of a change in plasma cholesterol.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: change (%) compared to baseline
Arm/Group | Cholic Acid
Number analyzed (Participants) | 12
change (%) compared to baseline | 37.8 (22.4)
Statistical Analysis 1: Comparison: Cholic Acid; Test type: Superiority; p = 0.011, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Cholic Acid
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
No limitations or caveats.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT03720990/Prot_SAP_000.pdf